CLINICAL TRIAL: NCT06889233
Title: MOTOR PROFICIENCY IN RELATION TO COGNITIVE FUNCTIONS AND SEVERITY IN CHILDREN WITH AUTISM SPECTRUM DISORDERS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Ali Abdelmoniem, senior physiotherapist, Cairo University
Other Study IDs: P.T.REC/012/005056
Record Dates: First submitted 2025-02-27; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder
Keywords: AUTISM; ASD; RAVEN; CARS; BOT2; FINE MOTOR SKILLS; Gross motor skills
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- observational group: We will assess cognitive function using the Raven's Progressive Matrices and measure the severity of autism using the Childhood Autism Rating Scale (CARS). These assessments will then be compared with the children's fine and gross motor abilities using BOT2 .
  Interventions: Behavioral: measuring cognitive functions, severity of autism , gross and fine motor skills

INTERVENTIONS:
Behavioral: measuring cognitive functions, severity of autism , gross and fine motor skills — measuring cognitive functions by RAVEN measuring severity by CARS measuring fine and gross motor functions by BOT2

SUMMARY:
To investigate the relationship between cognitive function, the severity of autism spectrum disorder (ASD), and the development of fine and gross motor skills in children with ASD

DETAILED DESCRIPTION:
A sample of 64 children with autism aged from 5 to 12 years recruited from centres and schools of special needs for intellectual and developmental disabilities to measure cognitive function using the Raven's Progressive Matrices and measure the severity of autism using the Childhood Autism Rating Scale (CARS). These assessments will then be compared with the children's fine and gross motor abilities

ELIGIBILITY:
Inclusion criteria:

1. Children had been diagnosed with ASD.
2. Their chronological age ranged from 5 years to 12 years.
3. Intelligence quotient (IQ) ranged from 55 to 85.

Exclusion criteria:

Any child with the following criteria would be directly excluded from the evaluation for the consistency of the sample and statistically obtained results:

1. The child with ASD and other motor disabilities.
2. Visual or hearing impairment.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: autistic children age ranged from 5 to 12 years
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
measuring motor proficiency (gross & fine motor skills ) by using BOT2 scale | 12 weeks

SECONDARY OUTCOMES:
measuring cognitive functions by RAVEN Progressive matrices | 12 weeks
  this scale items like puzzle and the child must extract the missed part from six choices

OTHER OUTCOMES:
measuring severity of autism by using CARS scale | 12 weeks
  this scale like questionnaire consisted of 15 question and parents or teacher give answers to this questions

CONTACTS AND LOCATIONS:
Overall Officials: Heba Kamal professor, professor of physical therapy, Study Chair — Cairo University; Alaa fahmy hassan El Nemer, lecturer of physical therapy, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy cairo university, Cairo, Dokki, Egypt